CLINICAL TRIAL: NCT01115712
Title: A Randomized Clinical Trial to Measure the Effect of Pioglitazone on Insulin Sensitivity in Healthy Overweight and Obese Males
Brief Title: Effects of Pioglitazone on Insulin Sensitivity in Healthy Overweight and Obese Males (MK-0000-170)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-170; 170 (Other: Merck)
Record Dates: First submitted 2010-04-30; First posted 2010-05-04 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Healthy; Overweight; Obesity
Keywords: Healthy Volunteers
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Pioglitazone 30 mg (Active Comparator): Pioglitazone 30 mg
  Interventions: Drug: Comparator: Pioglitazone; Drug: Comparator: Hyperinsulinemic Euglycemic Clamp
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo; Drug: Comparator: Hyperinsulinemic Euglycemic Clamp

INTERVENTIONS:
Drug: Placebo — Placebo (to match pioglitazone 30 mg) once daily
  Arms: Placebo
Drug: Comparator: Pioglitazone — Pioglitazone 30 mg once daily
  Arms: Pioglitazone 30 mg
Drug: Comparator: Hyperinsulinemic Euglycemic Clamp — Infusion of Glucose (20% dextrose) to achieve a glucose concentration of 90mg/dL; Infusion of Insulin at a rate of 10 mU/m2/minute from 0 to 180 minutes and at a rate of 40 mU/m2/minute from 180 to 360 minutes; Saline infusion at 60 minutes before the insulin and glucose infusions to keep the antecubital vein open.

SUMMARY:
The purpose of this study is to evaluate whether 30 mg of pioglitazone administered once daily for up to 28 days to healthy overweight and obese subjects will lead to a significant change in insulin sensitivity, measured in the setting of a hyperinsulinemic euglycemic clamp

ELIGIBILITY:
Inclusion Criteria:

* Subject has a BMI of greater than 28 kg/m^2 and less than or equal to 38 kg/m^2
* Subject has been a nonsmoker and/or has not used nicotine or nicotine-containing products for at least approximately 6 months
* Subject is willing to avoid major dietary changes for the duration of the study

Exclusion Criteria:

* Subject has history of diabetes (Type 1, Type 2 or steroid-induced)
* Subject has a history of hypersensitivity to pioglitazone or other thiazolidinediones
* Subject has a history of liver disease, other than non-alcoholic fatty liver disease or non-alcoholic steatohepatitis
* Subject has a history of congestive heart failure
* Subject has a active or past history of atherosclerotic heart disease, heart failure, osteoporosis, osteopenia, recurrent bone fractures, or anemia
* Subject has a history of stroke, chronic seizures, or major neurological disorder
* Subject has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological or renal abnormalities or diseases
* Subject has a history of neoplastic disease within the past 5 years

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glucose infusion rate (M) during the high dose portion of the hyperinsulinemic euglycemic clamp after 28 days of dosing. | Baseline and 28 days
Change from baseline in glucose infusion rate (M) during the high dose portion of the hyperinsulinemic euglycemic clamp after 14 days of dosing | Baseline and 14 days

SECONDARY OUTCOMES:
Change from baseline in glucose infusion rate (M) during the low dose portion of the hyperinsulinemic euglycemic clamp after 28 days of dosing. | Baseline and 28 days
Change from baseline in glucose infusion rate (M) during the low dose portion of the hyperinsulinemic euglycemic clamp after 14 days of dosing | Baseline and 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Shankar SS, Shankar RR, Railkar RA, Beals CR, Steinberg HO, Kelley DE. Early Clinical Detection of Pharmacologic Response in Insulin Action in a Nondiabetic Insulin-Resistant Population. Curr Ther Res Clin Exp. 2015 Aug 14;77:83-9. doi: 10.1016/j.curtheres.2015.08.001. eCollection 2015 Dec. PMID 26543510